CLINICAL TRIAL: NCT01935544
Title: Effectiveness of Two Techniques in Injection Site Spotting for Botulinum Toxin Injections: Echography or Electro Stimulation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHU-0153
Record Dates: First submitted 2013-05-06; First posted 2013-09-05 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Stroke
Keywords: Botulinum Toxin; Ultrasound-guidance; Stroke; Spasticity; Ultrasonography; Hemiplegia
MeSH Terms: conditions — Stroke; Muscle Spasticity; Hemiplegia

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- botulinum toxin injections (Experimental): The main objective is to compare the efficiency of botulinum toxin injections depending on the localization technique: ultrasound vs. electrical stimulation.
  Interventions: Device: Botulinum toxin injection
- ultrasound guidance (Other): The secondary objective is to demonstrate less painful localization associated to ultrasound-guidance
  Interventions: Device: Botulinum toxin injection

INTERVENTIONS:
Device: Botulinum toxin injection

SUMMARY:
Botulinum toxin injections are an effective treatment of limb spasticity after stroke. Different tracking techniques are used to locate a proper injection spot. Palpatory technique is barely effective and induces a high risk of error. Localization by electro stimulation is frequently used in adults, but often requires multiple painful repositioning of the needle. Ultrasound tracking is sometimes used in children but not much in adults.

The advantages of ultrasound-guided botulinum toxin injections are a painless localization and greater injection accuracy. Safety is therefore enhanced since intravascular injection is easily avoided.

The few existing publications on the subject are essentially case reports. Few studies have focused on comparing different injection techniques and so far, no well-conducted study has highlighted superior efficiency of ultrasound-guided injections.

DETAILED DESCRIPTION:
Objectives:

The main objective is to compare the efficiency of botulinum toxin injections depending on the localization technique: ultrasound vs. electrical stimulation.

The secondary objective is to demonstrate less painful localization associated to ultrasound-guidance.

Evaluations:

The primary endpoint is the variation of passive range of motion of ankle dorsiflexion at slow speed and high speed ("Tardieu scale") while keeping knee straight.

The secondary endpoints are:

* The other components of the "Tardieu scale": quality of muscle reaction (X) at slow speed and fast speed, angle of apparition of the muscle reaction (Y) at slow speed and fast speed.
* Assessment of spasticity of the triceps surae on the modified Ashworth scale.
* The walking speed.
* The extent of pain at the injection site by visual analogue scale.
* The duration of tracking and injection.

Methodology:

This prospective, randomized, single-center, single-blind, cross-over, study will be conducted in chronic stroke patients with spasticity of the triceps surae.

Patients will receive two injections during the protocol, each with a different technique of localization. Randomization will determine which technique will be used in the first and the second place.

Patients will be selected from the cohort of patients supported by consultation of Physical Medicine and Rehabilitation Department of the University Hospital of Clermont-Ferrand. Injections of botulinum toxin and assessments will take place in the same department.

The study period is five months for each patient. This study does not present a major risk for the subjects. The main inconvenience is injection pain or side effects of botulinum toxin (increase of motor deficits or dysphagia).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years.
* Hemiplegia sequelae of stroke
* Spasticity of the triceps surae listed at least 1 + / 4 on the modified Ashworth scale
* Ability to give written consent

Exclusion Criteria:

* Injection of botulinum toxin older than 3 months
* Patient who has already received ultrasound-guided injection of botulinum toxin
* Indication of botulinum toxin injection in other muscle groups in the lower limb than triceps surae
* Swallowing impairment
* Ongoing AVK anticoagulation treatment with INR greater than 3 during one week before randomization.
* Ongoing treatment by aminoglycosides
* General anesthesia with injection of curare planned during the participation in the protocol
* Wearing a pacemaker
* History of ankle arthrodesis
* Other cons-indication for botulinum toxin injection: myasthenia gravis, pregnancy, lactation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-11-19 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
Passive range of motion of ankle dorsiflexion (Tardieu scale) while keeping knee straight | at inclusion
Passive range of motion of ankle dorsiflexion (Tardieu scale) while keeping knee straight | at day 1 (first injection)
Passive range of motion of ankle dorsiflexion (Tardieu scale) while keeping knee straight | at day 60
Passive range of motion of ankle dorsiflexion (Tardieu scale) while keeping knee straight | at day 120 (second injection)
Passive range of motion of ankle dorsiflexion (Tardieu scale) while keeping knee straight | at day 150

SECONDARY OUTCOMES:
Tardieu scale: quality of muscle reaction at slow speed and fast speed | at Inclusion, D1, D60, D120 and D150
Angle of apparition of the muscle reaction at slow speed and fast speed | at Inclusion, D1, D60, D120 and D150
Spasticity of the triceps surae on the modified Ashworth scale | at Inclusion, D1, D60, D120 and D150
Walking speed | at Inclusion, D1, D60, D120 and D150
Extent of pain at the injection site by visual analogue scale | at D1, D120
Duration of tracking and injection | at D1, D120

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle HAURET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Morel C, Hauret I, Andant N, Bonnin A, Pereira B, Coudeyre E. Efficacy of two injection-site localisation techniques for botulinum toxin injections: a single-blind, crossover, randomised trial protocol among adults with hemiplegia due to stroke. BMJ Open. 2016 Nov 15;6(11):e011751. doi: 10.1136/bmjopen-2016-011751. PMID 27852706